CLINICAL TRIAL: NCT02720666
Title: K-001 Treatment of Advanced Pancreatic Cancer: Phase I Clinical Trial of Monotherapy's Tolerability
Brief Title: K-001 Treatment of Advanced Pancreatic Cancer: Clinical Trial of Monotherapy's Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Liwei Wang, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPOG001_01
Record Dates: First submitted 2016-02-13; First posted 2016-03-28 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A:K-001 2700mg/d (1350mg BID) (Experimental): K-001 1350mg twice a day, to be taken with warm water on an empty stomach; 4 weeks' administration for each group.
  Interventions: Drug: K-001
- Group B: K-001 3240mg/d (1620mg BID) (Experimental): K-001 1620mg twice a day, to be taken with warm water on an empty stomach; 4 weeks' administration for each group.
  Interventions: Drug: K-001
- Group C: K-001 3780mg/d (1890mg BID) (Experimental): K-001 1890mg twice a day, to be taken with warm water on an empty stomach; 4 weeks' administration for each group.
  Interventions: Drug: K-001
- Group D: K-001 4320mg/d (2160mg BID) (Experimental): K-001 2160mg twice a day, to be taken with warm water on an empty stomach; 4 weeks' administration for each group.
  Interventions: Drug: K-001

INTERVENTIONS:
Drug: K-001 — In case of severe adverse reactions associated with the test drug, or if half of the participants show adverse reactions at Ⅲ level and above, the test should be terminated. The maximum dosage not causing the above-described situation shall be considered as the maximum tolerated dose or the biologically effective dose. After the test, continuous medication shall be given upon request from patients.
  Other Names: Peptidoglycan Complex of Spirulina

SUMMARY:
This study is an open and single-center Phase I clinical research on patients with advanced pancreatic cancer, for evaluating their adverse reactions or tolerance to K-001, so as to determine the safe and reasonable dosage and dosing regimen.

DETAILED DESCRIPTION:
According to past experience to toxicology studies and clinical test, K-001 at a dose of 2700mg/day has a good safety profile for human body. Upon observation, pancreatic cancer patients receiving a medication at 2160mg/day (1080mg BID) have had good therapeutic efficacy, no sign of significant toxicity.

Dosing regimen:

Phase I clinical test: maximum dose of monotherapy at 2700mg/day. Four groups of repeated administration of monotherapy, at least 3 patients for each group.

Group A: 2700mg/d (1350mg BID); Group B: 3240mg/d (1620mg BID); Group C: 3780mg/d (1890mg BID); Group D: 4320mg/d (2160mg BID). Twice a day, to be taken with warm water on an empty stomach; 4 weeks' administration for each group.

In case of severe adverse reactions associated with the test drug, or if half of the participants show adverse reactions at Ⅲ level and above, the test should be terminated. The maximum dosage not causing the above-described situation shall be considered as the maximum tolerated dose or the biologically effective dose. After the test, continuous medication shall be given upon request from patients.

ELIGIBILITY:
Inclusion Criteria:

Disease-related criteria for inclusion:

1. Based on histodiagnosis or cytodiagnosis;
2. Locally advanced or metastatic pancreatic adenocarcinoma;
3. Failure of standard treatment, >28 days after the last chemotherapy;
4. Patients not suitable for or having given up standard treatment;
5. At least one lesion measurable according to RECIST V 1.0 criteria;
6. ECOG score: 0～1;
7. Expected survival: ≥3 months;

   Haematological, biochemical and organ functions:
8. Hematological indices:

   * Absolute neutrophil count: ≥1.5×109/L;
   * Platelet count: ≥80×109/L;
   * Hemoglobin: ≥9.0 g/dL.
9. Total bilirubin: ≤1.5 x ULN, albumin: ≥3.0g/dL;
10. Patients without liver metastasis: ALT (SGPT) & AST (SGOT) ≤3.0 x ULN Patients with liver metastasis: ALT (SGPT) & AST (SGOT)≤5.0 x ULN;
11. Renal functions: serum creatinine ≤ 1.5xULN, Ccr ≥ 60ml/min (Cockcroft-Gault);

    General criteria for inclusion:
12. Age: 18～70;
13. Letter of Consent signed by the patient or his/her legal representative:
14. Women of childbearing age must have a urine pregnancy test within 7 days before starting treatment, only negative results shall be included in the group. Male and female patients of childbearing age have agreed to use a reliable method of contraception before and during participating the study as well as 90 days (at least) after withdrawal.

Exclusion Criteria:

Disease-related criteria for exclusion:

1. Patients of pancreatic tumor but not adenocarcinoma;
2. Having received radiotherapy for his/her target lesions prior to this study, with no progress;
3. Known presence of brain metastases or leptomeningeal metastases;
4. With Vater's ampulla cancer or bile duct cancer;
5. Partial or complete intestinal obstruction;
6. History of other malignancies in past five years, except for:

   * A consecutive 5-year disease-free survival from single surgery of other malignancies;
   * Cured basal cell carcinoma and cured cervical carcinoma in situ.

   General criteria for exclusion:
7. Pregnant or breast-feeding women;
8. Any unstable systemic disease, including: active infection; hypertension uncontrollable by medication (≥160/100mmHg); unstable angina, or angina with the onset from within the last three months; congestive heart failure (≥level II according to New York Heart Association [NYHA], see Annex 4); myocardial infarction occurred within 1 year before the enrollment; severe arrhythmias requiring medical treatment; and mental disorders, etc.;
9. Presence of active hepatitis B (history of hepatitis B infection, whether with or without medication, HBV DNA≥104 copy number or ≥2000u/ml) or HCV-Ab positive; known HIV-positive patients (no clinical signs or symptoms suggesting exemption of HIV test for HIV-infected individuals);
10. Having received any of the following treatment within specific time period before inclusion:

    * Having had a major surgery within 4 weeks before inclusion;
    * Having received expanded scope of radiotherapy within 4 weeks, or having received limited scope of radiotherapy within 2 weeks before inclusion;
    * Having participated in any other therapeutic/interventive clinical trials within 4 weeks before inclusion, or taking part in an ongoing trial.
11. With CTCAE toxicity at level II or above (excluding hair loss or skin pigmentation), uncured and caused by any previous treatment;
12. Not fitting in the study, as conceived by the researcher.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) of K-001 | day 29
  The maximum-tolerated dose (MTD) of K-001 will be defined as the maximum dose level at which no more than one patient out of three experiences a dose-limiting toxicity (DLT) using Common Terminology Criteria for Adverse Events (CTCAE) criteria, version 4.0. If none of the patient experiences DLT, the maximum dose in the trial (4320mg/d) will be defined as MTD and the biologically effective dose.

SECONDARY OUTCOMES:
Change of life quality assessed using EORTC QLQ-C30 V 3.0 | within 7 days before taking drugs and day 8, day 15, day 22 and day 29
  EORTC QLQ-C30 V 3.0
Change from Baseline of the Treg cell count | within 14 days before taking drugs, day 15 and day 29
  Laboratory tests: blood immunity test of FOXP3+CD4+Treg cell count
Evaluation of suffered pains assessed using Numerical Rating Scale (NRS) | within 7 days before taking drugs and day 8, day 15, day 22 and day 29
  Numerical Rating Scale (NRS)
Change from Baseline of the C-reactive protein (CRP) | within 14 days before taking drugs, day 15 and day 29
  Evaluation the level of CRP with laboratory tests of blood.
Clinical efficacy of K-001 assessed by disease control rate (DCR) according to RECIST V 1.0 criteria | day 29
  Evaluate patients with imaging, including CT/MRI of the chest, abdomen and pelvic, and get disease control rate (DCR) according to RECIST V 1.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Xingpeng Wang, MD, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cui J, Yang H, Liu J, Chen D, Hu J, Zhang H, Wang Y, Han T, Mao T, Jiao F, Biskup E, Pan Y, Liu M, Wang L. A phase I study of the safety and activity of K-001 in patients with advanced pancreatic ductal adenocarcinoma. BMC Cancer. 2021 Jun 7;21(1):672. doi: 10.1186/s12885-021-08375-6. PMID 34098895